CLINICAL TRIAL: NCT04919330
Title: Embodying a Compassionate Self Through Acceptance and Commitment Therapy for Parents and Children With Eczema: A Family Based Eczema Management Programme
Brief Title: Acceptance and Commitment Therapy-based Eczema Management Programme
Acronym: ACTeczema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Yuen Yu CHONG, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RG2019/2020_A_7
Record Dates: First submitted 2021-06-04; First posted 2021-06-09 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Eczema
Keywords: Acceptance and Commitment Therapy; Eczema; Randomised Controlled Trial
MeSH Terms: conditions — Eczema

STUDY DESIGN:
Intervention Model Description: Parallel Assignment; repeated-measures 2-arm randomized controlled trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors and researchers (and health care staff of the study hospital) are blind to the group assignment and intervention undertaken and concealed to the participant list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ACT Group (Experimental): One four weekly 2-hour sessions of family ACT-based eczema management programme (FACT-EMP) and routine eczema care provided by the study hospital, including medical follow-ups and nurses' consultation.
  Interventions: Behavioral: Family Acceptance and Commitment Therapy-based Eczema Management Programme
- Wait-list Control Group (Other): Routine eczema care provided by the study hospital, including medical follow-ups and nurses' consultation
  Interventions: Behavioral: Wait-list Control Group

INTERVENTIONS:
Behavioral: Family Acceptance and Commitment Therapy-based Eczema Management Programme — The parent-child dyads will receive four weekly 2-hour sessions of family ACT-based eczema management programme (FACT-EMP). In each session, a group of 6-8 parent-child dyads will receive 90 minutes of ACT, followed by 30 minutes of education related to eczema management. Throughout the sessions, ACT strategies will help the dyads achieve the following therapeutic processes: To weaken the rumination cycle and "fused thoughts" related to eczema with body-image concern, shame and self-criticism for extending kindness and understanding to oneself; to build self-perspective-taking when seeing one's experience as part of the larger human experience; to strengthen their stands for their values related to self-kindness with acceptance of one's experience; and to take steps to act on values while practising kindness and compassion. Same as the waitlist control, the dyads will receive routine eczema care provided by the study hospital, including medical follow-ups and nurses' consultation.
  Arms: ACT Group
Behavioral: Wait-list Control Group — The parent-child dyads will receive routine eczema care provided by the study hospital, including medical follow-ups and nurses' consultation. To ensure equity of access to potentially effective treatment (i.e., family ACT-based eczema management programme), the dyads in the wait-list control group will receive the same programme after the completion of all assessments of the intervention arm.
  Arms: Wait-list Control Group

SUMMARY:
This pilot randomised wait-list controlled trial aims to determine the feasibility, acceptability and preliminary effects of a Family Acceptance and Commitment Therapy-based Eczema Management Programme (FACT-EMP) on the health outcomes of both children patients and their main caregivers over a 3-month post-intervention.

DETAILED DESCRIPTION:
Background:

Eczema is the most common paediatric skin condition affecting 15-20% children worldwide and 30% of children in Hong Kong. The highly visible nature of eczema symptoms that deviate from the individual's idealized body image could compromise his/her sense of self, leading to feelings of body image disturbance. It has been reported that children may use their illness to avoid schools, experience low self-esteem, shame and guilt and even stigmatization. In addition, their parents experience high level of stress in caring for their children with eczema, can easily generate shame and guilt feelings if they perceive themselves not performing satisfactory parenting roles in safeguarding their child's health. One emerging therapeutic approach to managing body-image concern, psychological difficulties associated with self-criticism and shame is by fostering self-compassion.

This study is a pilot randomized controlled trial aiming at examining the effects of a family-based eczema management programme in Hong Kong utilizing Acceptance and Commitment Therapy (ACT) to foster self-compassion of parents and their children affected by eczema. It is expected that fostering self-compassion could empower the parent-child dyads in cultivating a more loving, kind and forgiving attitude towards eczema, leading to improved motivation for self-care and better health outcomes. If found effective, the programme can improve the lives of many local families with children living with eczema through addressing their unmet psychological needs. In addition, the programme can be incorporated into current service in hospitals and community settings in Hong Kong and other Chinese communities.

Aim and hypothesis to be tested:

The proposed study will use a single-blinded, pilot randomized wait-list controlled trial design to determine the feasibility, acceptability and preliminary effects of a family ACT-based eczema management programme (FACT-EMP) on the health outcomes of both parent caregivers and children with eczema over 3-month post-intervention. It is hypothesized that when compared with a wait-list control group receiving standard care, the participants of the programme can show significant improvements in:

1. childhood eczema severity (primary outcome for children),
2. parental eczema management (primary outcome for parents),
3. parental depression, anxiety and stress,
4. health-related quality of life, psychological flexibility and self-compassion of both caregivers and their children with eczema immediately at immediately and 3-month post-intervention.

Design: A randomized wait-list controlled trial

Participants: Parents and their children aged 6-12 years diagnosed with eczema

Intervention condition: The parent-child dyads will receive four weekly 2-hour sessions of FACT-EMP. In each session, a group of 7-8 parent-child dyads will receive 90 minutes of ACT, followed by 30 minutes of education related to eczema management. The dyads in the wait-list control group will be offered to receive the same intervention after the completion of all assessments of the intervention arm.

Outcomes: The primary outcome for children is childhood eczema severity, while the primary outcome for parents is parental eczema management. The secondary outcomes for children are quality of life, self-compassion and psychological flexibility, while the secondary outcomes for parents are symptoms of depression, anxiety and stress, quality of life, psychological flexibility and self-compassion. The assessments of the aforementioned outcomes will be conducted at baseline, at post-intervention and at 3-month post-intervention by trained nurses/ research staff blinded to treatment allocation.

ELIGIBILITY:
Inclusion criteria:

The parent-child dyads should fulfil the following criteria:

1. For the child, he or she should be 6-12 years old and diagnosed with eczema by a physician as documented in the medical records.
2. For the parent, he or she should be 19-65 years; either father/mother in each family who is the primary caregiver responsible for the daily care of his/her child (e.g. the same parent who accompanied the child for follow-up appointments of the study hospital at every time), living together with the target child, able to communicate in Cantonese and accessible by telephone.

Exclusion criteria:

1. Any parent and/or his/her child who are currently participating in another eczema-related intervention study, or where the child has significant medical morbidities, including congenital problems, oxygen-dependent conditions, or the presence of tracheotomy, will be excluded.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2021-07-03 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Child's eczema severity | Change from baseline to 3 months post-intervention
  The Severity scoring of atopic dermatitis (SCORAD) will be used to assess the severity of childhood eczema, including the extent and intensity of the disease, and the degree of itching and sleep disturbance (Rehal et al., 2011).
Parent's self-efficacy of eczema management | Change from baseline to 3 months post-intervention
  The 29-item Chinese Version of Parental Self-Efficacy with Eczema Care Index (PASECI; Cheng et al., 2020) will be adopted to assess the parents' self-efficacy for performing eczema management tasks, managing the child's symptoms and behavior. The PASECI is arranged in 4 subscales: Managing Medication, Managing Eczema and Symptoms, Communicating with Health Professionals, and Managing Personal Challenges. Each item is scored on an 11-point Linkert scale, ranging from 0 (Cannot do at all) to 10 (Highly certain can do it). The scores of PASECI are gained by adding items up. The higher the PASECI score, the greater the parental self-efficacy in respective scales. The PASECI possessed high internal consistency (α=.97), test-retest reliability (ICC =.93-.99), and acceptable convergent validity in the Hong Kong population.

SECONDARY OUTCOMES:
Child's quality of life | Change from baseline to 3 months post-intervention
  The 10-item Children's Dermatology Life Quality Index (CDLQI; Chuh, 2003) will be used to assess the quality of life of children living with eczema. A total of six dimensions will be assessed comprising Symptoms and Feelings, Leisure, School or Holidays, Personal Relationships, Sleep, and Treatment. A 4-point scale is used, ranging from 0 (Not at all) to 3 (Very much/Prevented school). The 10-item CDLQI score is calculated by summing the scores of the 10 questions, giving a maximum of 30 and a minimum of 0. The higher the score, the greater the degree of handicap (the more quality of life is impaired). The CDLQI has high internal consistency and a strong correlation with physical-rated disease severity.
Child's self-compassion | Change from baseline to 3 months post-intervention
  The 12-item Self-Compassion Scale for Children (SCS-C; Sutton et al., 2018) will be adopted to measure the self-compassion of children. A 5-point scale is used, ranging from 1 (Never) to 5 (Always). Items on the Self-Compassion Scale for Children (SCS-C) addressed each of the six components of Neff's definition of self-compassion. The items assessing self-judgment, isolation, and over-identification were reverse-scored. The SCS-C comprises negatively-worded items and positively-worded items, each with acceptable internal consistency (α = .81-.83).
Child's psychological flexibility | Change from baseline to 3 months post-intervention
  The 10-item Child and Adolescent Mindfulness Measure (CAMM; Greco et al., 2011) will be adopted to measure the psychological flexibility in terms of acceptance and mindfulness of the children with a 5-point Linkert scale, ranging from 0 (Never true) to 4 (Always true). Total scores on the CAMM were computed by summing the responses to the 10 items, yielding a possible range of 0 - 40. The CAMM has good reliability (α = .78-.83) and positive correlations with quality of life, social skills, and academic performance as well as negative correlations with somatic complaints, internalizing and externalizing symptoms.
Parent's symptoms of depression, anxiety and stress | Change from baseline to 3 months post-intervention
  The 21-item Depression Anxiety Stress Scales-21 (DASS-21; Lovibond et al., 1995) will be applied to evaluate the parents' states of depression, anxiety, and stress. A 4-point Linkert scale is used, ranging from 0 (Did not apply to me at all) to 3 (Applied to me very much/most of the time) with 3 subscales consisting of Depression, Anxiety, and Stress. Higher scores indicate more frequent symptomatology. The reliabilities for the depression, anxiety, and stress subscales in the DASS-21 were .82, .88, and .90, respectively.
Parent's quality of life. | Change from baseline to 3 months post-intervention
  The 28-item Parents' Index of Quality of Life in Atopic Dermatitis (PIQoL-AD; McKenna et al., 2005) will be used to assess the quality of life of parents in caring for children with eczema with a dichotomous yes/no response format, 0 = No and 1 = Yes. The total score of PIQoL-AD ranging from 0 to 28, and a high score indicates poor quality of life. The PiQoL-AD is a standardized measure possessing good internal consistency (α=.88-.93) and test-retest reliability(r=.85) in various populations.
Parent's psychological flexibility | Change from baseline to 3 months post-intervention
  The 7-item Chinese version of the Acceptance and Action Questionnaire-II (AAQ-II; Chong et al., 2019) will be used to assess the psychological flexibility of the parents with a 7-point Likert scale, ranging from 1 (Never true) to 7 (Always true). The item scores are added together to create a total score (range 7 to 49). The higher the total score, the poor psychological flexibility (more psychologically inflexible), and the lower the total score, the better the psychological flexibility. The AAQ-II possessed good internal consistencies (α=.88) and test-retest reliabilities (r=.79-.81) in Hong Kong parents of children with asthma.
Parent's self-compassion | Change from baseline to 3 months post-intervention
  The 26-item Self Compassion Scale (SCS; Chen et al., 2011; Neff et al., 2016) will be adopted to measure self-compassion of the parents covering six domains: Self-Kindness, Self-Judgment, Common Humanity, Isolation, Mindfulness, and Over-Identification. An overall self-compassion score was calculated for each participant by reverse coding responses to the negatively worded items comprising self-judgment, isolation, and over-identification subscales, then calculating the means for each of the six subscales, and finally summing the means to create a total self-compassion score. The SCS has good internal reliability in Chinese and Western populations (α ≥ 0.86 in all samples).

CONTACTS AND LOCATIONS:
Overall Officials: Yuen Yu CHONG, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Paediatrics and Adolescent Medicine, Tuen Mun Hospital, Tuenmen, New Territories, Hong Kong

REFERENCES:
- [Derived] Chong YY, Chien WT, Mou HY, Leung SP, Wong OY, Lam SY. Acceptance and Commitment Therapy Eczema Management Program for Children With Eczema: A Pilot Randomised Controlled Trial. Clin Exp Allergy. 2025 Aug;55(8):701-715. doi: 10.1111/cea.70003. Epub 2025 Feb 3. PMID 39900107